CLINICAL TRIAL: NCT04635865
Title: Computer-Assisted Jaw Reconstruction Using 3D-Printed Patient-Specific Surgical Plates Versus Conventional Surgical Plates: A Randomised Controlled Clinical Trial
Brief Title: 3D-Printed Patient-Specific Surgical Plates Versus Conventional Surgical Plates in Jaw Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yuxiong Su, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-548
Record Dates: First submitted 2020-10-29; First posted 2020-11-19 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Mandibular Neoplasms; Maxillary Neoplasms; Dentofacial Deformities
Keywords: 3D printing; patient-specific titanium plate; mandibular malignancy; dento-maxillofacial deformity; mandibular reconstruction; maxillary reconstruction
MeSH Terms: conditions — Mandibular Neoplasms; Maxillary Neoplasms; Dentofacial Deformities

STUDY DESIGN:
Intervention Model Description: Patients fulfilling the eligibility criteria and willing to participate will be randomised after baseline assessment (1:1 allocation ratio). A priori, an independent statistician will prepare a computer-generated randomisation schedule in a random-sized permuted blocks of four or six patients stratified by location of reconstruction (maxilla/mandible) and gender (F/M) to ensure that the numbers of participants receiving the two interventions are closely balanced within each stratum. The allocation numbers will be concealed in opaque sealed envelopes prepared by a central study coordinator, only opening them after informed consent and baseline measures have been obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed patient-specific plate group (Experimental): 3D-printed patient-specific plate will be used for reconstruction in this patient group
  Interventions: Device: 3D-printed patient-specific plate
- Conventional plate group (Active Comparator): conventional commercial plates will be used for reconstruction in this patient group
  Interventions: Device: Conventional commercial reconstruction plate

INTERVENTIONS:
Device: 3D-printed patient-specific plate — We adopt an in-house approach for designing by surgeons. All patient-specific devices are designed in 3-matic 13.0 (Materialise). Both cutting and transferring guides are then additively manufactured by Fused Deposition Manufacturing (FDM) using ULTEM 1010, or by Stereolithography using MED610 resin (Stratasys Ltd, Eden Prairie, MN, USA). Both ULTEM 1010 and MED610 are FDA cleared biocompatible materials applicable to high-temperature autoclaving.
  Patient-specific surgical plates are designed by delineating a plate path on bone surface, then followed by the placement of screw holes. Surgical plates are generated by the built-in command in 3-matic. After that, surgical plates are fabricated by SLM using grade 2 titanium powder.
  Arms: 3D-printed patient-specific plate group
Device: Conventional commercial reconstruction plate — Bone segments will be stabilized using commercial titanium surgical plates (DePuy Synthes, United States), which are bent manually before fastening the screws.[
  Arms: Conventional plate group

SUMMARY:
Objectives: The aim of this randomised controlled clinical trial is to evaluate surgical accuracy and efficiency of computer-assisted jaw reconstruction using 3D-printed patient-specific titanium surgical plates versus conventional plates.

Hypothesis to be tested: The investigators hypothesize that compared to conventional surgical plates, 3D-printed patient-specific surgical plates improve surgical accuracy and efficiency of computer assisted jaw reconstruction.

Design and subjects: This is an open-label, prospective, double-arm, and single-centre randomised controlled clinical trial. Patients with maxillary or mandibular neoplastic, inflammatory and congenital diseases who require immediate or secondary reconstructive surgery will be invited to participate in the study.

Study instruments: 3D-printed patient-specific titanium surgical plates and conventional plates.

Main Outcome Measures: The primary endpoint is the accuracy of reconstruction. The secondary endpoints include the accuracy of osteotomy, reconstruction time, total operative time, intraoperative blood loss, length of post-operative hospital stay, and postoperative adverse events.

Data analysis: The accuracy parameters, reconstruction time, total operative time, intraoperative blood loss, length of post-operative hospital stay will be presented as mean values with standard deviations. The post-operative adverse events will be calculated and presented as frequency with standard deviation.

Expected results: This randomised control trial will prove improved accuracy and efficiency of reconstruction using 3D printed patient-specific titanium surgical plates. This study is expected to provide high-level evidence to push forward the popularity of using 3D medical printing technology in surgical field.

DETAILED DESCRIPTION:
This randomised controlled clinical trial was based on our previous clinical trial "Three-Dimensional Printing of Patient-Specific Titanium Plates in Jaw Surgery: A Pilot Study" (HKU/HA HKW IRB, No. UW 16-315; registered in ClinicalTrials.gov with a No. of NCT03057223; supported by HMRF Project no.: 05161626).

Over the past few decades, autologous vascularized bone flaps have become the preferred choice for head and neck reconstruction. The anastomosed blood supply endows vascularized bone flaps with improved survival rate and inherent anti-infection performance. Along with the development of microvascular surgery, surgeons are seeking more accurate reconstruction to enhance better aesthetic and functional outcomes. However, a main disadvantage of autologous bone flaps is the mismatch in the shape of donor bone, which need to be cut and trimmed to fit the defects and better restore the natural appearance. Much efforts have been devoted to facilitate bone manipulations, and then the computer-assisted surgery (CAS) emerged in the 21st century as a viable option. In CAS, surgeons do virtual plans in computer, which then guide the precise harvest and arrangement of bone segments for repairing defects in the operating theatre. Bone segments can be fine-navigated to best restore the original skeleton. In previous researches, various devices have been developed to navigate bone segments according to virtual plans, including cutting templates, skull models, and surgical navigation system.

However, the missing link between bone navigation and accurate reconstruction is the plate fixation procedure. In a conventional manner, bone segments are fixed using commercial off-the-shelf titanium plates, which should be manually bent and twisted to fit bone anatomy. The manual contouring process is often tedious and technique-demanding, and adversely affect the precise location of bone segments. What's worse, repeated bending can even lead to poor fatigue performance. The disadvantages of conventional surgical plates make it necessary to develop patient-specific surgical plates. Compared to conventional plates, patient-specific surgical plates are designed and manufactured in 3D structures aligned with individual bone contours. Instead of contouring plates based on anatomical structure of bones in conventional plates, patient-specific surgical plates navigate the folding and precise location of bone segments, and hopefully improve the accuracy of reconstruction. Meanwhile, since no plate bending is required, patient-specific surgical plates can be used to optimize bone reconstruction in a more efficient and standardized manner.

In recent years, with the rapid development of additive manufacturing (3D printing), it is now feasible to manufacture patient-specific metal implants with topologically optimized structures. Many efforts have been made to develop porous bone scaffolds for regenerative medicine, which are endowed with customized porosity to achieve optimal biomechanical properties. However, although additively manufactured bone scaffolds demonstrate excellent performance in some complicated cases, they still cannot replace the dominant role of autologous vascularized bone flaps in head and neck reconstruction. Therefore, it is of crucial importance to explore the application of additive manufactured (3D printed) patient-specific surgical plates, albeit not much research has been done in this direction.

In our previous study (HKU/HA HKW IRB, No. UW 16-315) supported by Health and Medical Research Fund (Project no.: 05161626), the investigators have successfully manufactured patient-specific titanium plates with high precision through selective laser melting (SLM) technology, which is a high-tech 3D printing technology that fully melts titanium powders into complete entities in the layer by layer manner. SLM enables the fabrication of patient-specific titanium surgical plates with tailored structures and outstanding biomechanical properties. Our results showed promising clinical outcomes in the application of 3D printed patient-specific titanium plates in head and neck reconstruction. Furthermore, the investigators did a retrospective study comparing the patients who had undergone jaw reconstructive surgery using 3D printed patient-specific surgical plates versus conventional titanium plates and the result showed superior accuracy of reconstruction outcomes in the study group with the use of 3D printed patient-specific surgical plates. However, there were significant limitations in our study. First, as a retrospective study, the innate flaw of study design was unavoidable, such as selection bias. Second, there was significantly difference in follow-up periods between the study group and control group. The imaging data used for accuracy analysis were obtained during different post-operative periods, which compromised the final outcomes. Finally, surgical efficiency endpoints, such as operation time, blood loss, and post-operative hospital stay, which could be significantly affected by multiple confounding factors, are difficult to control by retrospective study design. Hence, there is still lack of high-level evidence concerning the advantages of 3D printed patient-specific surgical plates in head and neck reconstruction. Whether 3D printed patient-specific surgical plates improve surgical accuracy and efficiency compared to conventional plates in computer assisted jaw reconstruction should be further investigated before large-scale clinical application.

Therefore, the investigators aim to evaluate surgical accuracy and efficiency of computer-assisted jaw reconstruction using 3D-printed patient-specific titanium surgical plates versus conventional plates in a prospective randomised controlled clinical trial. Our study is expected to provide high-level evidence to push forward the popularity of using 3D medical printing new technology in the surgical field.

Methods

The methodology has already been set up and has been proved feasible in our earlier studies. The PI has been working on computer aided surgical simulation, virtual planning, and 3D printed surgical templates in the maxillofacial surgery for several years and has published a series of articles.

1. Computer-assisted Surgery

   The CAS techniques used in head and neck reconstruction are well established in our unit and have been described previously. Briefly, CAS is composed of three main phases: the pre-operative phase of the virtual surgery and 3D printing of patient-specific devices, intra-operative phase involving precision-enhanced surgery to install the patient-specific devices, and post-operative phase involving the accuracy analysis. The patient-specific devices can include cutting guides, positioning guides, and the patient-specific titanium plates. In our trial, the study group will use cutting guides and patient-specific titanium plates, whereas the control group will use cutting guides, positioning guides, and conventional plates.

   In the pre-operative phase, the virtual surgery will be performed by surgeons using the ProPlan CMF 2.0 software (Materialise, Leuven, Belgium). The patient's CT data is initially segmented to rebuild 3D virtual models of the maxilla or mandible using ProPlan's interactive interface. Next, bone resection is performed in the 3D models for en bloc removal of any tumours. Meanwhile, bone grafts are harvested from fibula or iliac crest to repair defects and restore the normal appearance. Finally, the virtually reconstructed maxilla or mandible is used to design patient-specific devices to navigate the bone segments.
2. Additive Manufacturing of Patient-specific Devices

   Compared to the conventional approach of designing patient-specific devices using engineering companies, we have adopt an in-house approach that allow the surgeons to design and manufacture the devices. All patient-specific devices are designed in 3-matic 13.0 (Materialise). Cutting guides, which guide and adapt to bone surface for accurate bone resection, are generated by wrapping to the bone surface.

   For the study group, patient-specific surgical plates are designed by delineating the plate path on the bone surface, followed by the placement of screw holes. Surgical plates are generated by a built-in command in 3-matic. Next, the surgical plates are fabricated by SLM using grade 2 titanium powder. For the control group, positioning guides will be designed for the bone segment alignment and inset.

   Both cutting and positioning guides will be additively manufactured by Fused Deposition Manufacturing (FDM) using ULTEM 1010, or by Stereolithography using MED610 resin (Stratasys Ltd, Eden Prairie, MN, USA). Both ULTEM 1010 and MED610 are FDA cleared biocompatible materials usable in high-temperature autoclaving.
3. Surgical Procedures

   In the present study, all patients in both groups will undergo CAS carried out by the same chief surgeon (PI). During the surgery, patient-specific cutting guides will enable precise jawbone resection and bone flap osteotomy.

   In the control group, the arrangement of bone segments will be manipulated according to the positioning guide. Bone segments will be stabilized using commercial titanium surgical plates (DePuy Synthes, United States), which are bent manually before fastening with screws. In the study group, patient-specific surgical plates will be designed and fabricated to custom-fit the bone contours of reconstructed maxilla or mandible. The screw holes embedded in cutting guides correspond to the 3D-printed patient-specific surgical plates, which will guide the position of surgical plates and bone segments, thereby facilitating folding, positioning, and fixation of bone segments in the real surgery. Standard peri-operative management will be similar in both groups. Post-operative follow-up will be conducted in a routine manner.
4. Data collection procedures

CT scan will be obtained at baseline (before surgery) and post-operatively (within 1 month after the surgery). The accuracy of reconstruction will be independently assessed by two assessors. Training will be provided using previous cases, and calibration between the two assessors will be done with the aim of achieving over 90% inter-assessor agreement in three consecutive training cases before starting the measurement of subject cases in this study. Other information such as reconstruction time, total operative time, intra-operative blood loss, length of post-operative hospital stay, and post-operative adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, of both gender;
* Provision of signed and dated informed consent form;
* Diagnosed with maxillofacial benign or malignant tumours or inflammatory or congenital diseases and indicated for computer-assisted jaw surgery;
* Primary or secondary reconstruction with autogenous bony free flaps or graft will be needed;
* Titanium plates will be used for internal fixation for the reconstruction surgery;
* Agree to comply with follow-up procedures.

Exclusion Criteria:

* Patients who are pregnant;
* Patients who have medically compromised conditions and cannot tolerate the surgery;
* Systemic conditions or diseases that violate the normal bone healing;
* Patients who are unable to take the preoperative and postoperative CT/CBCT scans;
* Patients who are unable to have a two-week period prior to surgery, for virtual surgery simulation, 3D patient-specific surgical plate design and fabrication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Accuracy of reconstruction | through study completion, an average of 5 years
  The primary endpoint is accuracy of reconstruction, which is defined as the distance or angulation deviations of anatomical landmarks between the virtual plan and actual surgical outcome.

SECONDARY OUTCOMES:
accuracy of osteotomy | after surgery for each case, through study completion, an average of 5 years
  Deviation of actual osteotomy from the digital planning
reconstruction time | during surgery for each case, through study completion, an average of 5 years
  time from the start of flap ischemia to the finish of anastomosis and internal fixation
total operative time | during surgery for each case, through study completion, an average of 5 years
  total operative time
intraoperative blood loss | during surgery for each case, through study completion, an average of 5 years
  intraoperative blood loss
length of post-operative hospital stay | after surgery for each case, through study completion, an average of 5 years
  length of post-operative hospital stay
postoperative adverse events | after surgery for each case, through study completion, an average of 5 years
  postoperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiong Su, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- The Prince Philip Dental Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rifkin WJ, Kantar RS, Ali-Khan S, Plana NM, Diaz-Siso JR, Tsakiris M, Rodriguez ED. Facial Disfigurement and Identity: A Review of the Literature and Implications for Facial Transplantation. AMA J Ethics. 2018 Apr 1;20(4):309-323. doi: 10.1001/journalofethics.2018.20.4.peer1-1804. PMID 29671724
- [Background] Lang H, France E, Williams B, Humphris G, Wells M. The psychological experience of living with head and neck cancer: a systematic review and meta-synthesis. Psychooncology. 2013 Dec;22(12):2648-63. doi: 10.1002/pon.3343. Epub 2013 Jul 10. PMID 23840037
- [Background] Hanasono MM, Matros E, Disa JJ. Important aspects of head and neck reconstruction. Plast Reconstr Surg. 2014 Dec;134(6):968e-980e. doi: 10.1097/PRS.0000000000000722. PMID 25415120
- [Background] Hurvitz KA, Kobayashi M, Evans GRD. Current options in head and neck reconstruction. Plast Reconstr Surg. 2006 Oct;118(5):122e-133e. doi: 10.1097/01.prs.0000237094.58891.fb. PMID 17016169
- [Background] Powcharoen W, Yang WF, Yan Li K, Zhu W, Su YX. Computer-Assisted versus Conventional Freehand Mandibular Reconstruction with Fibula Free Flap: A Systematic Review and Meta-Analysis. Plast Reconstr Surg. 2019 Dec;144(6):1417-1428. doi: 10.1097/PRS.0000000000006261. PMID 31764662
- [Background] Yang WF, Choi WS, Leung YY, Curtin JP, Du R, Zhang CY, Chen XS, Su YX. Three-dimensional printing of patient-specific surgical plates in head and neck reconstruction: A prospective pilot study. Oral Oncol. 2018 Mar;78:31-36. doi: 10.1016/j.oraloncology.2018.01.005. Epub 2018 Jan 16. PMID 29496055
- [Background] Takizawa T, Nakayama N, Haniu H, Aoki K, Okamoto M, Nomura H, Tanaka M, Sobajima A, Yoshida K, Kamanaka T, Ajima K, Oishi A, Kuroda C, Ishida H, Okano S, Kobayashi S, Kato H, Saito N. Titanium Fiber Plates for Bone Tissue Repair. Adv Mater. 2018 Jan;30(4). doi: 10.1002/adma.201703608. Epub 2017 Dec 7. PMID 29215204
- [Background] Ciocca L, Mazzoni S, Fantini M, Persiani F, Marchetti C, Scotti R. CAD/CAM guided secondary mandibular reconstruction of a discontinuity defect after ablative cancer surgery. J Craniomaxillofac Surg. 2012 Dec;40(8):e511-5. doi: 10.1016/j.jcms.2012.03.015. Epub 2012 Apr 30. PMID 22551671
- [Background] Wang X, Xu S, Zhou S, Xu W, Leary M, Choong P, Qian M, Brandt M, Xie YM. Topological design and additive manufacturing of porous metals for bone scaffolds and orthopaedic implants: A review. Biomaterials. 2016 Mar;83:127-41. doi: 10.1016/j.biomaterials.2016.01.012. Epub 2016 Jan 6. PMID 26773669
- [Background] Karageorgiou V, Kaplan D. Porosity of 3D biomaterial scaffolds and osteogenesis. Biomaterials. 2005 Sep;26(27):5474-91. doi: 10.1016/j.biomaterials.2005.02.002. PMID 15860204
- [Background] van Hengel IAJ, Riool M, Fratila-Apachitei LE, Witte-Bouma J, Farrell E, Zadpoor AA, Zaat SAJ, Apachitei I. Selective laser melting porous metallic implants with immobilized silver nanoparticles kill and prevent biofilm formation by methicillin-resistant Staphylococcus aureus. Biomaterials. 2017 Sep;140:1-15. doi: 10.1016/j.biomaterials.2017.02.030. Epub 2017 Feb 28. PMID 28622569
- [Background] Shaoki A, Xu JY, Sun H, Chen XS, Ouyang J, Zhuang XM, Deng FL. Osseointegration of three-dimensional designed titanium implants manufactured by selective laser melting. Biofabrication. 2016 Oct 27;8(4):045014. doi: 10.1088/1758-5090/8/4/045014. PMID 27788123
- [Background] Xu JY, Chen XS, Zhang CY, Liu Y, Wang J, Deng FL. Improved bioactivity of selective laser melting titanium: Surface modification with micro-/nano-textured hierarchical topography and bone regeneration performance evaluation. Mater Sci Eng C Mater Biol Appl. 2016 Nov 1;68:229-240. doi: 10.1016/j.msec.2016.05.096. Epub 2016 May 24. PMID 27524017
- [Background] Yang WF, Choi WS, Wong MC, Powcharoen W, Zhu WY, Tsoi JK, Chow M, Kwok KW, Su YX. Three-Dimensionally Printed Patient-Specific Surgical Plates Increase Accuracy of Oncologic Head and Neck Reconstruction Versus Conventional Surgical Plates: A Comparative Study. Ann Surg Oncol. 2021 Jan;28(1):363-375. doi: 10.1245/s10434-020-08732-y. Epub 2020 Jun 22. PMID 32572853